CLINICAL TRIAL: NCT03153527
Title: Glucocorticoid Withdrawal and Glucocorticoid-induced Adrenal Insufficiency: a Randomized Controlled Multicenter Trial
Brief Title: Taper Or Abrupt Steroid Stop: TOASSTtrial
Acronym: TOASST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Baselland Bruderholz (Other); Swiss National Science Foundation (Other); HEMMI Stiftung Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-00487; ex14Rutishauser
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Disorder; Autoimmune
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Standard treatment arm: Prednisone, a synthetic glucocorticoid with intermediate duration of action (biological half-life 18-35 hrs). The detailed characteristics of the compound, marketed under several brand names, can be found at www.swissmedicinfo.ch: Prednison Streuli (Swissmedic registration number: 29349); Prednison Axapharm (Swissmedic registration number: 58761); Prednison Galepharm (Swissmedic registration number: 50821).
  Interventional treatment arm: matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding of trial participants, treating physicians, study doctors, study nurses, outcome assessors and data analysts will be ensured by using identical-looking placebo, packaged in identical vials as the prednisone verum. Vials will be labeled with "Prednisone or Placebo" in an identical fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo arm (intervention arm) (Placebo Comparator): Stop glucocorticoid treatment; administer placebo matching the verum preparation in weekly intervals.
  Interventions: Other: Placebo Arm
- Verum group (control/standard arm) (Active Comparator): If patient is on > 7.5 mg prednisone-equivalent daily: administer 7.5 mg q.d. for 7 days, then 5 mg q.d. for 7 days, then 2.5 mg q.d. for 7 days, then 2.5 mg q.d. every second day, then stop. If patient on 7.5 mg q.d.: maintain for 7 days, then taper as above.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — The control intervention (standard treatment) consists of prednisone treatment in decreasing doses, starting with 7.5 mg q.d. and reducing the dose every 7 days, such that prednisone treatment is stopped after a total of 4 weeks.
  Arms: Verum group (control/standard arm)
Other: Placebo Arm — The experimental intervention consists of stopping glucocorticoid treatment abruptly and administering matching placebo over 4 weeks.
  Arms: Placebo arm (intervention arm)

SUMMARY:
This study is an Investigator-initiated, placebo-controlled, multicenter noninferiority trial, comparing rapid termination of systemic glucocorticoid treatment with a tapering regime over 4 weeks.

DETAILED DESCRIPTION:
In total, 573 patients will be enrolled. Patients will be randomly assigned in a 1:1 ratio to either prednisone in decreasing doses over 4 weeks or placebo.

Patients, treating physicians, and study personnel will be blinded to treatment allocation to either prednisone or matching placebo. At inclusion, we will perform a 250 micrograms Synacthen® stimulation test. The results of the test will be blinded to treating physicians and investigators, and its value to predict clinical outcome will only be assessed after completion of the trial. As a safety measure, all patients will be instructed about stress coverage as well as signs and symptoms of hypocortisolism and will be provided with emergency medication. Patients will be randomized to the standard (tapering) or the experimental (matching placebo) arm. Follow-up will be for six months. In order to improve adherence to the study and ensure feasibility, follow-up visits in most study centers will be by telephone only. Visits will be performed early after stopping glucocorticoids in both arms (i.e. at days 7 and 35) to ensure safety; the other two visits will be on days 90 and 180.

Amendment approved in 1-2018: former exclusion criterion 'status post organ transplantation' was revised and deleted

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age ≥ 18 years
* Daily glucocorticoid dose ≥ 7.5 mg prednisone-equivalent at the time of inclusion
* Therapy over ≥ 28 days, ≥ 7.5 mg average daily dose, with a cumulative glucocorticoid dose ≥ 420 mg prednisone-equivalent prior to inclusion
* Tapering not or no longer mandatory to treat underlying disease

Exclusion Criteria:

* Primary adrenal failure
* Treatment with systemic depot glucocorticoids (e.g. intramuscular, epidural)
* Incapability to administer glucocorticoid cover treatment in situations of stress
* Inability or unwillingness to provide informed consent
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to any incidence | up to 6 months
  Time to first occurrence of hospitalization, death, initiation of unplanned systemic glucocorticoid therapy, or adrenal crisis (defined as glucocorticoid-responsive hypotension or shock with or without accompanying symptoms and signs such as weakness, apathy, nausea, vomiting, abdominal pain, hypothermia, hyponatremia [serum sodium < 135 millimole (mM)], hyperkalemia [serum potassium > 5 mM], hypoglycemia [plasma glucose < 3.5 mM]); whichever occurs first.

SECONDARY OUTCOMES:
Time to specific incidence | up to 6 months
  Time to first occurrence of individual components of the primary outcome;
Cumulative overall systemic glucocorticoid dose | up to 6 months
  Cumulative overall systemic glucocorticoid dose
Cumulative systemic glucocorticoid dose administered to treat or prevent adrenal failure | up to 6 months
  Cumulative systemic glucocorticoid dose administered to treat or prevent adrenal failure
Cumulative systemic glucocorticoid dose administered to treat relapse | up to 6 months
  Cumulative systemic glucocorticoid dose administered to treat relapse of disease, specified for each disease
General health status | assessed at days 1, 7, 28, 35, 90,180
  General health status as self-assessed by the participant on a visual analog scale (VAS) from 0 to 100
Score of symptoms and signs of hypocortisolism | up to 6 months
  Score of symptoms and signs of hypocortisolism: weakness, hypothermia, nausea, vomiting, abdominal pain, fatigue, dizziness, Blood pressure, serum Na and serum glucose concentrations.
Performance in 250 mcg Synacthen® test | up to 6 months
  Performance in 250 mcg Synacthen® test: test assessed day 1 in all participants, plus days 7 and 35 in those followed in centers Bruderholz, Luzern, Aarau
In patients hospitalized at study entry: length of hospital stay | up to 6 months
  In patients hospitalized at study entry: length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Rutishauser, Prof MD, Principal Investigator — Departement Medizin, Kantonsspital Baden
Locations (15):
- Germany (2):
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Würzburg, Würzburg
- Switzerland (13):
  - Departement of Internal Medicine, Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Endocrinology/Diabetology/Metabolism; University Hospital Basel, Basel
  - Department of Rheumatology, Immunology, and Allergology, Inselspital, Bern
  - Division of Gastroenterology, Spital Bülach AG, Bülach
  - Kantonsspital Frauenfeld, Frauenfeld
  - Geneva University Hospitals, Geneva
  - Center for Primary Health Care,University of Basel, Kantonsspital Baselland, Liestal
  - Internal Medicine, Kantonsspital Baselland/Liestal, Liestal
  - Department of Internal Medicine, Kantonsspital Münsterlingen, Münsterlingen
  - Stoffwechselzentrum, Kantonsspital Olten, Olten
  - Department of Internal Medicine, Kantonsspital St. Gallen, Sankt Gallen
  - Dept. of Endocrinology, Diabetology and Clinical Nutrition, University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No
No sharing planned

REFERENCES:
- [Derived] Komminoth M, Donath MY, Hepprich M, Schuetz P, Blum CA, Mueller B, Reny JL, Gosselin P, Breville G, Brandle M, Henzen C, Leuppi JD, Kistler AD, Thurnheer R, Beuschlein F, Rudofsky G, Aeberli D, Villiger PM, Bohm S, Chifu I, Fassnacht M, Meyer G, Bojunga J, Cattaneo M, Sluka C, Schneider H, Rutishauser J; <<TOASST>> study group. Glucocorticoid withdrawal and glucocorticoid-induced adrenal insufficiency: Study protocol of the randomized controlled <<TOASST" (Taper Or Abrupt Steroid STop) multicenter trial. PLoS One. 2023 Apr 5;18(4):e0281585. doi: 10.1371/journal.pone.0281585. eCollection 2023. PMID 37018188